CLINICAL TRIAL: NCT05208255
Title: Investigation of the Effect of Telerehabilitation-Based Exercise and Motor Imagery Training on ADHD Symptoms, and Balance in Children With ADHD: A Pilot Study
Brief Title: Effect of Telerehabilitation-Based Exercise and Motor Imagery Training in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Nurullah Buker, Research asisstant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Buker N
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Adhd
Keywords: ADHD; Telerehabilitation; Motor Imagery; Balance; Physiotherapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group1 (Experimental): The telerehabilitation-based neurocognitive exercise group
  6 weeks, 2 sessions per week Session duration: 60 minutes
  Interventions: Other: Exercise
- Exercise Group2 (Experimental): The telerehabilitation-based neurocognitive exercise+motor imagery training group
  6 weeks, 2 sessions per week Session duration: 60 minutes (45 minutes-neurocognitive exercise; 15 minutes-motor imagery training)
  Interventions: Other: Exercise
- Control Group (Active Comparator): The medication group - Participants who voluntarily participated in the study but did not want to participate in exercise groups.
  6 weeks of medication use
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — NEP is a multimodal exercise program including different motor coordination exercises and cognitive tasks. Exercises are progressed from simple to complex tasks. Varied equipment (such as different sized balls, rackets, tulles, exercises balls, eye bands, ropes etc.) is used during different exercises containing cross-limb movements, throwing, jumping, walking, and cognitive tasks. Although the stages of the NEP and exercise selection are the same for each participant, the use of materials or cognitive tasks selection may differ according to the age and skill of the participant. The cognitive tasks were performed by using different visual (colored cards, numbered cards etc.) or auditory cues.
  Motor Imagery Program: Motor imagery (MI) is a dynamic mental state during which the representation of a given motor movement is rehearsed in working memory without overt motor output. MI training will be performed in the form of imagined NEP exercises in the last 15 minutes of the session.
  Other Names: Neurocognitive Exercise Program (NEP)

SUMMARY:
The study was prospectively planned and conducted as per protocol. However, registration was completed retrospectively due to administrative oversight. No changes were made to the protocol after study initiation.

Attention Deficit Hyperactivity Disorder (ADHD) is a common neurodevelopmental disorder characterized by inattention, hyperactivity, and impulsivity.

About one-third of children with ADHD have difficulties with fine and gross motor skills. Motor problems during dynamic balance tasks are more pronounced in these children compared to their typically developing peers. These issues may result from dysfunction in brain regions, possibly linked to delayed cerebellar development. Motor imagery-the mental simulation of movement without actual execution-has been studied as a cause of motor impairments in ADHD and Developmental Coordination Disorder (DCD). While motor imagery deficits are clear in DCD, evidence in ADHD remains unclear.

Studies show that motor imagery training, alone or combined with physical exercise, can improve postural control. In children with DCD, motor imagery training improved movement skills.

ADHD treatment is multidimensional, including pharmacological and psychosocial interventions. Medications are effective in reducing symptoms and associated behaviors. Physical exercise also helps reduce ADHD symptoms, improving medication response and cognitive functions.

This study aims to examine the effects of telerehabilitation-based exercise and motor imagery training on ADHD symptoms and balance in children. Telerehabilitation has become popular due to pandemic-related restrictions, yet no exercise program combining telerehabilitation and motor imagery exists for children with ADHD.

DETAILED DESCRIPTION:
The study was prospectively planned and conducted as per protocol. However, registration was completed retrospectively due to administrative oversight. No changes were made to the protocol after study initiation.

Attention Deficit Hyperactivity Disorder (ADHD) is one of the most common neurodevelopmental disorders in children. 7.2% in the world; ADHD with a prevalence of approximately 13% in Turkey; It is a disorder that affects impulsivity, inattention and hyperactivity symptoms, and affects daily life activities and causes inadequacies.

Children with ADHD have lower motor skills and performance than healthy children; reported to have higher motor coordination disorders. It has been shown that one-third of children with ADHD have problems with tasks that require fine and gross motor skills. In addition, it was stated that the motor skill problems experienced during dynamic situations were more pronounced than healthy children. It has been reported that motor disorders seen in children with ADHD may result from dysfunction in some related brain regions, and that especially delayed or impaired cerebellar development may contribute to the pathophysiology of ADHD. ADHD can cause significant academic, social and psychiatric problems. If left untreated, these problems continue for life.

Motor imagery was investigated as the underlying cause of motor impairment in children with ADHD and Developmental Coordination Disorder (DDD). It was stated that motor imagery was significantly impaired in children with ADHD. But this situation was not clear in children with ADHD. Motor imagery is defined as the mental thinking of a movement without actual movement being revealed. It has been reported that combined physical and motor imagery programs applied at different rates, as well as motor imagery training without physical exercise, are effective in improving postural control. In a study conducted with children with DCD, it was shown that motor imagery training improves children's movement skills.

In the treatment of ADHD, there are multidimensional treatment approaches that include medical and psychosocial interventions. Psychostimulants are the drugs most commonly used in the treatment of ADHD. Pharmacological treatments, including stimulant and non-stimulant drugs, are highly effective in reducing ADHD's attention deficit and hyperactivity/impulsivity features and associated destructive behaviors. In addition, from psycho-educational interventions; Multiple approach models that combine psychosocial intervention such as family education, school-oriented regulation, cognitive behavioral therapy, and social education have also been found to be effective methods. When looking at the effective exercise methods on ADHD symptoms, there are mostly studies on aerobic exercises and other physical exercises. Also, other physical exercises are known to reduce ADHD symptoms. It has been shown that exercise methods enable patients receiving drug therapy to respond better to drugs and improve cognitive functions in ADHD cases.

Due to the Coronavirus disease (Covid-19), which started in the last months of 2019 and whose negative effects are still continuing, some difficulties are experienced in the health systems. This situation has led to a greater tendency towards telerehabilitation applications during the treatment and follow-up process. Telerehabilitation is a method that aims to provide rehabilitation to patients and clinicians by using information and communication technologies by reducing obstacles such as distance, time and cost. Although telerehabilitation programs have been used in different disease groups in recent years, these programs use is not common in children with ADHD.

In conclusion, motor imagery disorder is unclear in children with ADHD. In addition, there are different opinions about the underlying aetiology of motor coordination and balance problems that cause children with ADHD to have difficulties in daily life and sports activities. The use of telerehabilitation methods has become widespread due to the difficulties in conducting face-to-face treatment and follow-up processes due to the pandemic. In addition, there is no exercise program based on telerehabilitation and motor imagery in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* Between the ages of 7-12
* Volunteer
* Not using psychostimulant drugs for at least two months

Exclusion Criteria:

* Having a systemic disease that affects physical assessments
* Having severe visual impairment (color blindness, strabismus, etc.)
* Having a neurological disease
* Having a musculoskeletal disease
* Having any neuropsychiatric disorder other than Oppositional Defiant Disorder, anxiety disorders, and mood disorders
* Having Developmental Coordination Disorder
* Have previously participated in a motor imaging or motor imaging-like study/practice
* Having an IQ score of 80 and below
* Being a licensed athlete

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Conners Parent Rating Scale-Revised Short | pre-intervention
  It determines the severity of ADHD symptoms. The scale consists of three sub-scales (Oppositional Defiant, Cognitive Problems-Inattention, Hyperactivity) and an auxiliary scale (ADHD Index). The questions are answered by the parents on a four-point Likert scale as "Never", "rarely", "often", and "always" which are scored as "0", "1", "2", and "3", respectively.
Conners Parent Rating Scale-Revised Short | within the first week post-intervention
  It determines the severity of ADHD symptoms. The scale consists of three sub-scales (Oppositional Defiant, Cognitive Problems-Inattention, Hyperactivity) and an auxiliary scale (ADHD Index). The questions are answered by the parents on a four-point Likert scale as "Never", "rarely", "often", and "always" which are scored as "0", "1", "2", and "3", respectively.
Stroop Test | pre-intervention
  The Stroop Test is a task assessing executive function involving processing speed, concentration, and selective attention. Stroop Test was applied in five sections. These sections and related cards are as follows in their application order: (1) The card with the color names printed in black (1st card); (2) the card with the color names printed in different colors (2nd card); (3) the card with the colored printed circles (3rd card); (4) in the card with neutral words without the color name (4th Card); (5) the section where the colors of the words in the 2nd Card are spelt, with the names of colors printed in different colors.
Stroop Test | within the first week post-intervention
  The Stroop Test is a task assessing executive function involving processing speed, concentration, and selective attention. Stroop Test was applied in five sections. These sections and related cards are as follows in their application order: (1) The card with the color names printed in black (1st card); (2) the card with the color names printed in different colors (2nd card); (3) the card with the colored printed circles (3rd card); (4) in the card with neutral words without the color name (4th Card); (5) the section where the colors of the words in the 2nd Card are spelt, with the names of colors printed in different colors.
d2 Test of Attention | pre-intervention
  The d2 Test measures processing speed, rule compliance, and quality of performance, allowing for a neuropsychological estimation of individual attention and concentration performance.
d2 Test of Attention | within the first week post-intervention
  The d2 Test measures processing speed, rule compliance, and quality of performance, allowing for a neuropsychological estimation of individual attention and concentration performance.
Y Balance Test | pre-intervention
  Y-Balance Test is used to evaluate the dynamic balance. YBT is performed in three directions (anterior, posteromedial, and posterolateral).
Y Balance Test | within the first week post-intervention
  Y-Balance Test is used to evaluate the dynamic balance. YBT is performed in three directions (anterior, posteromedial, and posterolateral).
Timed Up and Go Test | pre-intervention
  The Timed Up and Go Test, which is found an excellent level of validity and reproducibility by Nicolini and Donadio, is performed as the standard test protocol applied in children to evaluate dynamic balance and functionality.
Timed Up and Go Test | within the first week post-intervention
  The Timed Up and Go Test, which is found an excellent level of validity and reproducibility by Nicolini and Donadio, is performed as the standard test protocol applied in children to evaluate dynamic balance and functionality.

SECONDARY OUTCOMES:
Movement Imagery Questionnaire-Revised Second Edition | pre-intervention
  The Motion Imagery Questionnaire-Revised Second Edition will be used to measure children's visual and kinesthetic visualization skills. It consists of 14 items, seven of which are visual and 7 of which are kinesthetic. During the test, children scores by asking them to perform the actions in the instruction once in reality, then to visualize the movement they do and to indicate the clarity of this imagery on a Likert-type scale from 1 (Very difficult to feel/see) to 7 (Very easy to feel/see).
Movement Imagery Questionnaire-Revised Second Edition | within the first week post-intervention
  The Motion Imagery Questionnaire-Revised Second Edition will be used to measure children's visual and kinesthetic visualization skills. It consists of 14 items, seven of which are visual and 7 of which are kinesthetic. During the test, children scores by asking them to perform the actions in the instruction once in reality, then to visualize the movement they do and to indicate the clarity of this imagery on a Likert-type scale from 1 (Very difficult to feel/see) to 7 (Very easy to feel/see).
Kinesthetic and Visual Imagery Ouestionnaire | pre-intervention
  The form consists of a total of 10 movements that measure five visual and five kinesthetic visualization skills developed to determine the extent to which individuals visualize and feel the imagined movements. The evaluator performs the relevant move on himself and then asks the participant to do the same movement only once. Then, the participant imagines the movement, and the visual clarity of the imaged movement or the senses are scored with the help of a 5-point ordinal scale.
Kinesthetic and Visual Imagery Ouestionnaire | within the first week post-intervention
  The form consists of a total of 10 movements that measure five visual and five kinesthetic visualization skills developed to determine the extent to which individuals visualize and feel the imagined movements. The evaluator performs the relevant move on himself and then asks the participant to do the same movement only once. Then, the participant imagines the movement, and the visual clarity of the imaged movement or the senses are scored with the help of a 5-point ordinal scale.
Timed Up and Go-Mental Chronometer | pre-intervention
  This test will be performed while sitting position in a chair at the beginning of the Timed Get Up and Go Test track. Individuals are asked to complete the TUG by imagining with their eyes closed, and the time to complete the test is recorded with a chronometer. The temporal coherence between the real and the imagined movement is calculated in terms of delta time with the formula '(real motion-imagined motion) / [(real motion+imagined motion) / 2] x 100'.
Timed Up and Go-Mental Chronometer | within the first week post-intervention
  This test will be performed while sitting position in a chair at the beginning of the Timed Get Up and Go Test track. Individuals are asked to complete the TUG by imagining with their eyes closed, and the time to complete the test is recorded with a chronometer. The temporal coherence between the real and the imagined movement is calculated in terms of delta time with the formula '(real motion-imagined motion) / [(real motion+imagined motion) / 2] x 100'.
Ruler Drop Test | pre-intervention
  It is a simple and inexpensive test used to evaluate the hand reaction time. For the test, a 50 cm ruler will be used. During the test, the person is asked to sit comfortably with his dominant arm on the table. The practitioner randomly leaves the ruler at hand level for 2-5 seconds, and the person is asked to grasp the ruler as quickly as possible. The distance the person has caught the ruler is recorded. The average of three measurements made after two trial tests will be taken as the test value.
Ruler Drop Test | within the first week post-intervention
  It is a simple and inexpensive test used to evaluate the hand reaction time. For the test, a 50 cm ruler will be used. During the test, the person is asked to sit comfortably with his dominant arm on the table. The practitioner randomly leaves the ruler at hand level for 2-5 seconds, and the person is asked to grasp the ruler as quickly as possible. The distance the person has caught the ruler is recorded. The average of three measurements made after two trial tests will be taken as the test value.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No